CLINICAL TRIAL: NCT04617015
Title: Defining and Treating a New Pediatric Asthma Endotype: Depression-related Asthma Mediated by the Cholinergic Pathway
Brief Title: Defining and Treating Depression-related Asthma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Heather Lehman, Clinical Associate Professor of Pediatrics, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00000774; UL1TR001412 (NIH)
Record Dates: First submitted 2019-07-24; First posted 2020-11-05 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Asthma; Depression; Childhood Asthma
Keywords: asthma; depression; anticholinergic therapy
MeSH Terms: conditions — Asthma; Depression | interventions — Ipratropium

STUDY DESIGN:
Intervention Model Description: Children with asthma and depression versus children with asthma without depression are compared for presence of allergies, airway inflammation, and response to bronchodilation with ipratropium.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ipratropium bromide (Experimental): All subjects will receive ipratropium bromide HFA and will have spirometry performed before and after ipratropium.
  Interventions: Drug: Ipratropium Bromide

INTERVENTIONS:
Drug: Ipratropium Bromide — All subjects receive inhaled ipratropium once with measurement of spirometry before and after. Bronchodilator response of subjects with depression is compare to that of subjects without depression.

SUMMARY:
Depression is seen more often in people with asthma, and may lead to increased development and severity of asthma.

This study will investigate whether children with depression and asthma have less allergic disease and less inflammation than children with asthma who do not have symptoms of depression.

The study will also investigate whether the lungs of children with depression and asthma respond to an anticholinergic inhaler called ipratropium more than the lungs of non-depressed asthmatic children.

DETAILED DESCRIPTION:
It is well accepted that asthma is not a single uniform disease, but rather many different disease sub-entities with different etiologies and pathophysiologies. The term "endotype" was coined to delineate distinct subtypes of asthma; an "endotype" specifically is as "a subtype of a condition, which is defined by a distinct functional or pathophysiological mechanism". The division of asthma into endotypes is critical to the development of targeted immunomodulators and other specific treatment modalities to more effectively treat the diverse asthmatics encountered in clinical practice.

There is a clear association between depression and asthma, with evidence suggesting that depression leads to increased development of asthma rather than the reverse. If, as suggested, depression truly mediates a subset of asthma, this depression-related asthma "endotype" has not been well characterized to date. A promising theory of the pathophysiological mechanism of depression-related asthma is that of autonomic nervous system dysregulation associated with depression leading to airway compromise (Miller and Wood, 2003). Specifically, depression is associated with excess parasympathetic (cholinergic) activation, and cholinergic activation can mediate bronchoconstriction through the action of acetylcholine on the muscarinic receptors on bronchial smooth muscle. It has been demonstrated that during emotional stimuli, depressed children with asthma have increased parasympathetic activation, which associates with increased airway resistance. In contrast, when experiencing these same emotional stimuli, non-depressed children with asthma have increased sympathetic activation.

The investigators anticipate that depressed child asthmatics have cholinergically-mediated bronchoconstriction as a major mediator of their disease activity. Based upon studies of depressed asthmatic children showing increased parasympathetic/cholinergic reactivity in response to laboratory based emotional stimuli, along with a recent study showing that depressed asthmatic adults have decreased bronchodilatory response to beta-agonists, the investigators hypothesize that asthmatic children with higher depressive indices will have more bronchodilatory response on spirometry following treatment with a short-acting inhaled anticholinergic, and less additional bronchodilation with an inhaled beta-agonist, compared to children with lower depressive indices. The investigators will set out to demonstrate if during an episode of bronchoconstriction, depressed child asthmatics will achieve more bronchodilation from a short-acting inhaled anticholinergic than will non-depressed child asthmatics.

The investigators next predict that with excess cholinergic activation as a cause of bronchoconstriction in depressed pediatric asthmatics, there will be less atopic sensitization and Th2-mediated inflammation driving the airway disease in this subset of asthmatics. The investigators hypothesize that, compared to non-depressed child asthmatics, depressed pediatric asthmatics during an episode of bronchoconstriction will show less evidence of airway inflammation as measured by fractional exhaled nitric oxide (FeNO) and peripheral blood eosinophilia, and will have lower rates of atopic sensitization measured by skin prick testing to environmental allergens and/or elevated total serum immunoglobulin E (IgE). In addition, the investigators will assess patient-identified asthma triggers, which are anticipated to be different in the depressed asthmatic group, with increased identification of emotions and cold weather as triggers, and less identification of allergens as triggers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* Decreased lung volumes for age/height/race (FEV1 80% predicted or FEV1/FVC 85%) on day of study visit assessed by spirometry.

Exclusion Criteria:

* Severely developmentally delayed patients, or those who suffer from other severe cognitive impairment not allowing them to perform spirometry or participate in study instruments.
* Patients who are pregnant or nursing.
* Patients with significant cardiopulmonary disease other than asthma, including cystic fibrosis, alpha-1-antitrypsin deficiency, interstitial lung disease, tracheo-/bronchomalacia, or cyanotic congenital cardiac defect.
* Patients with glaucoma, myasthenia gravis, or bladder neck obstruction (anticholinergics can worsen these conditions).
* Patients currently taking another anticholinergic medication

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
FEV1 percent change post-ipratropium | 30 minutes
  change in lung function measurement in response to anti-cholinergic medication

SECONDARY OUTCOMES:
FEV1 percent change post-albuterol | 15 minutes
  change in lung function measurement in response to beta-adrenergic medication
Number of positive environmental skin tests | 20 minutes
  Sensitization to environmental allergens measured by skin prick testing
ATI mood score | 5 minutes
  This score rates self-identified mood triggers of asthma on Asthma Trigger Inventory, an instrument used to assess self-perceived asthma triggers.
  The Asthma Trigger Inventory mood score ranges between 0 and 40 points. Higher score on the emotional trigger subscale indicated more self-perceived impact of emotions on asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Heather K Lehman, MD, Principal Investigator — SUNY at Buffalo School of Medicine and Biomedical Sciences
Locations (1):
- Women and Children's Hospital of Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No